CLINICAL TRIAL: NCT05439915
Title: Pilot Study of Asthma Diagnosis Through Peak Flows
Brief Title: Asthma Diagnosis Through Peak Flows
Acronym: DAPF-CSL
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Consorci Sanitari de Terrassa (Other)
Responsible Party: Principal Investigator, Joan Torras Borrell, Family Medicine, Principal Investigator, Clinical mentor, Consorci Sanitari de Terrassa
Other Study IDs: 02-22-161-062
Record Dates: First submitted 2022-06-27; First posted 2022-06-30 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Asthma
Keywords: asthma - diagnosis; maximal expiratory flow rate
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The guidelines indicate the possibility of diagnosing asthma through peak flow. This recommendation being the result of expert consensus, but the evidence is limited and contradictory. The aim of the present study is to assess whether the diagnosis of asthma through peak flow is not inferior to that of spirometry with bronchodilator test, which is the gold standard test. This is a pilot study to validate a diagnostic test. Its location is an urban health centre (CAP Sant Llàtzer of the Consorci Sanitari de Terrassa). Participation will be offered to all adult patients (18 years of age or older) who are suspected of having an asthma diagnosis. On the one hand, the reversibility will be determined by performing the peak flow test in the center with the administration of 4 puffs of salbutamol. On the other hand, PBD spirometry will be performed to complete the study and diagnosis of the patient. Peak flow is faster, cheaper, simpler, more accessible and safer for professionals in the context of an airbone pandemic.

DETAILED DESCRIPTION:
The pandemic has had a strong impact on healthcare quality standards in Catalonia. Prioritization at the primary level of immediate care over scheduled care has led to a decrease in continuity in patient care.

Asthma is a common treatable disease and exacerbations are preventable with proper staging and treatment if necessary. During the present pandemic, the ability to diagnose it through the test of choice (spirometry with bronchodilator test) has been compromised, taking into account the risks arising for health personnel to perform. This fact has conditioned that in the pandemic context it is recommended to limit its use as much as possible.

These reasons led to the suspension of spirometry at the beginning of the pandemic and later, although they have been restarted with the indicated filters to improve safety for patients and professionals, it has not been possible to restore normally for issues arising from the care pressure associated with the pandemic.

When the investigators reviewed the clinical guidelines, they specify that the diagnosis of asthma can also be made by measuring the maximum expiratory flow (PEF) with the peak flow. The measurement of PEF is simple, objective, non-invasive, and adds value to daily clinical practice, helping to define severity and contributing to patient self-management of the disease. The guidelines recommend that the diagnosis through peak flow is a degree of evidence C as the studies are very small samples and therefore the recommendation is based more on the consensus of experts than on the studies available.

However, these guidelines propose two alternative techniques: variability and reversibility.

The first is to measure with the peak flow of the daily variability of the maximum expiratory flow (PEF) in 2 weeks that would allow to diagnose asthma. But there is a difference in criteria in the variability of PEF per se between the two most frequently used guides in our environment.

On the one hand, according to the criteria in the Spanish Guide to Asthma Management (GEMA) the variability required for diagnosis must be greater than or equal to 20% in more than three days in a week for a two-week record. On the other hand, in the Global Initiative for Asthma (GINA) the diagnosis would be with a minimum variability of 10% in a single week, also monitored for a period of two weeks.

Both documents also explain the second technique: the possibility of using the reversibility of pre- and post-bronchodilation PEF with 4 Salbutamol poufs as a diagnostic tool. In this case, both guidelines agree that a reversibility greater than 20% would be a value to be taken into account in the diagnosis of asthma.

According to the available literature, the daily variability of PEF correlates better with bronchial hyperreactivity than with symptoms and airway obstruction, when used for monitoring asthmatic patients already known to have clinical stability. This variability provides information on the risk of exacerbations, and has long been recognized as a possible diagnostic tool (8).

Monitoring of PEF variability in children is insufficient to recommend this technique (9,10), although we must keep in mind that the diagnosis and monitoring of asthma in children is more difficult than in adults.

Other disadvantages of PEF should also be borne in mind: low reproducibility, lack of precise reference values in population groups and may underestimate airway obstruction. Some studies suggest that the usefulness of PEF for the diagnosis of asthma should be reconsidered despite what the guidelines recommend, while others recommend its use.

It is because of this need and the contradictions in the method and in the available evidence that the investigators propose to review patients who have pending spirometry with a suspected diagnosis of asthma and who have also not been able to perform them due to problems related to pandemic.

People with suspected asthma criteria will have a PEF test with a peak flow at the pre- and post-administration center of salbutamol to check the diagnosis for reversibility. In the pilot study, we do not plan to carry out peak flow controls at home for 14 days to assess variability in an attempt to keep it simpler, but we do consider a larger study with more centers depending on funding possibilities. The investigators will review these data if they can be correlated with the results of the same patients in a spirometry with bronchodilator test as this technique becomes available and it is possible to perform it safely for health personnel.

ELIGIBILITY:
Inclusion Criteria:

* Suspition of asthma, not yet confirmed.

Exclusion Criteria:

* No acceptance.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients visiting in an urban health centre with clinical suspition of asthma, not yet confirmed.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of asthma | 2 months
  Diagnosis of asthma through reversivility in peak flow compared to spirometry with bronchodilator test.

SECONDARY OUTCOMES:
Acceptation | 2 months
  Degree of acceptance of the patients with respect to the technique of the reversibility of the peak flows.
Ratios | 2 months
  To calculate the ratio of positive and negative likelihood for the reversibility of the peak flow
Sensitivity and specifity | 2 months
  To calculate the sensitivity and specificity for the reversibility of the peak flow with respect to spirometry with bronchodilator test.
Preference | 2 months
  To know the patients 'preference between spirometry with bronchodilator test and the reversibility of the peak flow.
Predisposition | 2 months
  To know the predisposition of patients to perform a study of variability with peak flows for 14 days.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coma E, Mora N, Mendez L, Benitez M, Hermosilla E, Fabregas M, Fina F, Mercade A, Flayeh S, Guiriguet C, Ballo E, Martinez Leon N, Mas A, Cordomi S, Lejardi Y, Medina M. Primary care in the time of COVID-19: monitoring the effect of the pandemic and the lockdown measures on 34 quality of care indicators calculated for 288 primary care practices covering about 6 million people in Catalonia. BMC Fam Pract. 2020 Oct 10;21(1):208. doi: 10.1186/s12875-020-01278-8. PMID 33038926
- [Background] Coma E, Mora N, Peremiquel-Trillas P, Benitez M, Mendez L, Mercade A, Fina F, Fabregas M, Medina M. Influence of organization and demographic characteristics of primary care practices on continuity of care: analysis of a retrospective cohort from 287 primary care practices covering about 6 million people in Catalonia. BMC Fam Pract. 2021 Mar 25;22(1):56. doi: 10.1186/s12875-021-01414-y. PMID 33761874
- [Background] Crimi C, Impellizzeri P, Campisi R, Nolasco S, Spanevello A, Crimi N. Practical considerations for spirometry during the COVID-19 outbreak: Literature review and insights. Pulmonology. 2021 Sep-Oct;27(5):438-447. doi: 10.1016/j.pulmoe.2020.07.011. Epub 2020 Aug 5. PMID 32800783
- [Background] Reddel HK, Salome CM, Peat JK, Woolcock AJ. Which index of peak expiratory flow is most useful in the management of stable asthma? Am J Respir Crit Care Med. 1995 May;151(5):1320-5. doi: 10.1164/ajrccm.151.5.7735580.
- [Background] Reddel HK, Taylor DR, Bateman ED, Boulet LP, Boushey HA, Busse WW, Casale TB, Chanez P, Enright PL, Gibson PG, de Jongste JC, Kerstjens HA, Lazarus SC, Levy ML, O'Byrne PM, Partridge MR, Pavord ID, Sears MR, Sterk PJ, Stoloff SW, Sullivan SD, Szefler SJ, Thomas MD, Wenzel SE; American Thoracic Society/European Respiratory Society Task Force on Asthma Control and Exacerbations. An official American Thoracic Society/European Respiratory Society statement: asthma control and exacerbations: standardizing endpoints for clinical asthma trials and clinical practice. Am J Respir Crit Care Med. 2009 Jul 1;180(1):59-99. doi: 10.1164/rccm.200801-060ST. PMID 19535666
- [Background] Hetzel MR, Clark TJ. Comparison of normal and asthmatic circadian rhythms in peak expiratory flow rate. Thorax. 1980 Oct;35(10):732-8. doi: 10.1136/thx.35.10.732. PMID 7466721
- [Background] Brouwer AF, Brand PL. Asthma education and monitoring: what has been shown to work. Paediatr Respir Rev. 2008 Sep;9(3):193-9; quiz 199-200. doi: 10.1016/j.prrv.2008.03.001. Epub 2008 Jul 30. PMID 18694711
- [Background] Sly PD, Landau LI, Weymouth R. Home recording of peak expiratory flow rates and perception of asthma. Am J Dis Child. 1985 May;139(5):479-82. doi: 10.1001/archpedi.1985.02140070053032. PMID 3984972
- [Background] Vaughan TR, Weber RW, Tipton WR, Nelson HS. Comparison of PEFR and FEV1 in patients with varying degrees of airway obstruction. Effect of modest altitude. Chest. 1989 Mar;95(3):558-62. doi: 10.1378/chest.95.3.558. PMID 2920583
- [Background] Goldstein MF, Veza BA, Dunsky EH, Dvorin DJ, Belecanech GA, Haralabatos IC. Comparisons of peak diurnal expiratory flow variation, postbronchodilator FEV(1) responses, and methacholine inhalation challenges in the evaluation of suspected asthma. Chest. 2001 Apr;119(4):1001-10. doi: 10.1378/chest.119.4.1001. PMID 11296161
- [Background] Jamison JP, McKinley RK. Validity of peak expiratory flow rate variability for the diagnosis of asthma. Clin Sci (Lond). 1993 Sep;85(3):367-71. doi: 10.1042/cs0850367. PMID 8403810
- [Background] Pignataro FS, Bonini M, Forgione A, Melandri S, Usmani OS. Asthma and gender: The female lung. Pharmacol Res. 2017 May;119:384-390. doi: 10.1016/j.phrs.2017.02.017. Epub 2017 Feb 24. PMID 28238829
- See also: GEMA 5.0. Guía española para el manejo del asma. Sociedad Española de Neumología y Cirugía Torácica, 2020. ISBN: 978-84-17372-97-2. — http://www.gemasma.com.
- See also: Global initiative for Asthma. Global Strategy for Asthma Management and Prevention, 2021. — http://www.ginasthma.org
- See also: Instituto Nacional de estadística. — http://www.ine.es/jaxiT3/Tabla.htm?t=7947
- See also: CIBERES: Centro de investigación biomédica en red de enfermedades respiratorias. — http://www.ciberes.org
- See also: Miquel-Gomara Perelló J, Román Rodríguez M. Medidor de Peak-flow: técnica de manejo y utilidad en Atención Primaria. MEDIFAM, 2002; 3: 206-213. — https://scielo.isciii.es/pdf/medif/v12n3/tecnicas.pdf